CLINICAL TRIAL: NCT00005522
Title: Social Dominance, Gender, and Cardiovascular Reactivity
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5049; R29HL058528 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-10

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Disease
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Coronary Disease

SUMMARY:
To examine biopsychosocial processes that might contribute to the associations among social dominance, gender, and cardiovascular reactivity,.

DETAILED DESCRIPTION:
BACKGROUND:

Social dominance, the tendency to exercise social influence and control, has been positively associated with coronary heart disease (CHD) risk among males, independent of biomedical risk factors and hostility. Exposure to dominant others behaviors also has been associated with elevated CHD risk. For females, submissiveness and a constellation of psychosocial behaviors opposite to urgency and competitiveness have been associated with increased risk for cardiovascular disease (CVD). The studies extend a growing literature concerning the central role of social relationships in health and illness and they test a theoretical model that addresses why social relationships and interpersonally-oriented person variables such as dominance may have differing consequences for the physical well-being of men and women.

DESIGN NARRATIVE:

The three studies were designed to test a social-contextual model of dominance and cardiovascular stress reactivity (CVR) that synthesized and elaborated earlier models in order to account for (1) cardiovascular consequences of exposure to dominant others and (2) differences in dominant men's and women's cardiovascular responses to social interactions. Because of the disproportionately high rates of CVD among Black Americans, both Black and white men and women were included in the studies.

Using a laboratory social interaction paradigm, study 1 refined and validated a coding system designed to assess dominant and hostile behaviors during dyadic social interaction. Study 2 examined two factors proposed to account for differences in dominant men's and women's cardiovascular responses to social interaction: (1) explicit role demands regarding dominance expression (i.e., the degree to which situations provided clear and salient cues regarding expected and acceptable behavior) and (2) gender composition of the dyad (i.e., same sex versus opposite sex). These two factors were manipulated independently while unacquainted, healthy young adult men and women participated in task-oriented dyadic discussions designed to activate motives to influence; cardiovascular responses were measured during the discussions and preceding rests. Study 3, a secondary analysis of data collected in study 2, examined associations between CVR and exposure to others' dominance. The aforementioned behavioral coding system was used to assess behavioral dominance observed in study 2 and path analytic techniques were used to model associations among CVR, one's own and one's partner's trait and behavioral dominance, gender, and situational factors.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1998-05; Study Completion 2004-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Newton — Boston University

REFERENCES:
- [Background] Kiecolt-Glaser JK, Newton TL. Marriage and health: his and hers. Psychol Bull. 2001 Jul;127(4):472-503. doi: 10.1037/0033-2909.127.4.472. PMID 11439708
- [Background] Newton TL, Philhower CL. Socioemotional correlates of self-reported menstrual cycle irregularity in premenopausal women. Psychosom Med. 2003 Nov-Dec;65(6):1065-9. doi: 10.1097/01.psy.0000097346.39776.59. PMID 14645787
- [Background] Newton TL, Watters CA, Philhower CL, Weigel RA. Cardiovascular reactivity during dyadic social interaction: the roles of gender and dominance. Int J Psychophysiol. 2005 Sep;57(3):219-28. doi: 10.1016/j.ijpsycho.2005.03.001. PMID 15882912